CLINICAL TRIAL: NCT03247998
Title: GASTROKE- the Effect of General Anesthesia Versus Sedation for Patients With Acute Ischemic STROKE Undergoing Endovascular Treatment on Three Month Morbidity and Mortality: a Feasibility Study.
Brief Title: GA vs. CS for Endovascular Stroke Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Miguel Arango, Anesthesiologist, Associate Professor, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GA Stroke
Record Dates: First submitted 2017-07-26; First posted 2017-08-14 (Actual); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Stroke; Endovascular Repair; Anesthesia
Keywords: Stroke; endovascular repair; general anesthesia; conscious sedation
MeSH Terms: conditions — Stroke | interventions — Anesthesia, General; Conscious Sedation; Remifentanil

STUDY DESIGN:
Intervention Model Description: There will be two arms of this study. In the first arm, the patients who meet the inclusion criteria of the study will be randomized to receive general anesthesia during endovascular treatment for stroke. In the second arm of the study, patients will receive general sedation during endovascular treatment.
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor who will analyze the outcome variables for this study (consciousness, motor function, sensation, speech, coordination, standard of care follow up assessments etc.) that may be impacted by choice of anesthesia/analgesia will be blinded to the treatment group of the participants to ensure unbiased reporting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia (Experimental): Patients who have had a stroke and meet the inclusion criteria for the study will receive general anesthesia during endovascular treatment. Choice of anesthetic for general anesthesia is dependent upon the patient condition and decision of the treating anesthesiologist (ketamine, propofol, fentanyl, midazolam,dexmedetomidine etc.). General Anesthesia Protocol: (Melinda J. Davis, Cynthia R. Campos-Herrera, & David P. Archer, 2012; Powers et al., 2015; Talke et al., 2014). Patient will be monitored in accordance with standard monitoring guidelines and the rest of the procedure will proceed in accordance with standard of care.
  See Detailed Description for additional details and description of follow-up procedures.
  Interventions: Drug: General Anesthesia
- Conscious Sedation with Remifentanil (Experimental): Patients who have had a stroke and meet the inclusion criteria for the study will receive conscious during endovascular treatment. Sedation will be accomplished using Remifentanil: 0.01-0.06 micrograms/kilogram/minute, titrated to effect. (Janssen et al., 2016). Patients who have had a stroke and meet the inclusion criteria for the study will receive general anesthesia during endovascular treatment. Patient will be monitored in accordance with standard monitoring guidelines and the rest of the procedure will proceed in accordance with standard of care.
  See Detailed Description for additional details and description of follow-up procedures.
  Interventions: Drug: Conscious Sedation with Remifentanil

INTERVENTIONS:
Drug: General Anesthesia — Patients who have had a stroke and meet the inclusion criteria for the study will receive general anesthesia during endovascular treatment. Choice of anesthetic for general anesthesia is dependent upon the patient condition and decision of the treating anesthesiologist (ketamine, propofol, fentanyl, midazolam,dexmedetomidine etc.). Induction of general anesthesia will follow standard treatment methods (Davis et al, 2012, Powers et al. 2015 Talke et al. 2015). Patient monitoring and care will proceed in accordance with standard of care guidelines. Refer to Detailed Description section for complete protocol information.
  Other Names: No other names
  Arms: General Anesthesia
Drug: Conscious Sedation with Remifentanil — Patients who have had a stroke and meet the inclusion criteria for the study will receive conscious during endovascular treatment. Sedation will be accomplished using Remifentanil: 0.01-0.06 micrograms/kilogram/minute, titrated to effect. (Janssen et al., 2016). Patient monitoring and care will proceed in accordance with standard of care guidelines. Refer to Detailed Description section for complete protocol information.
  Other Names: No other names
  Arms: Conscious Sedation with Remifentanil

SUMMARY:
After a stroke caused by a blockage (clot) in a blood vessel in the brain, patients may have the clot removed by threading a catheter from the groin up to the affected area of the brain. An anesthesiologist is involved in the patient's care during this procedure to maximize patient safety and procedural efficiency. The options for anesthesia for this procedure are general anesthesia (where the patient is unconscious) or sedation (where the patient is in a relaxed, calm, sleepy condition). Currently, it is unclear which of these anesthetic options contributes to the best patient outcome. The investigators would like to investigate whether or not one method of anesthesia (general or sedation) is better to use than the other when removing the clot.

DETAILED DESCRIPTION:
Rationale: Stroke is a leading cause of adult morbi-mortality worldwide. Intravenous (IV) recombinant tissue plasminogen activator (rtTPA) was the only therapeutic option for many years. After the publication of five randomized controlled trials, guidelines for stroke treatment were updated and released in 2015. According to these guidelines, in addition to IV rtTPA, endovascular therapy (EVT) for acute ischemic stroke (AIS), secondary to proximal intracranial arterial occlusion, has become established as an international standard of care (Avitsian & Machado, 2016). Management of patients undergoing stroke is complex due to the association of acute neurological physiological changes and pre-existing co-morbidities. To facilitate efficient and safe delivery of endovascular treatment, patients require anesthetic intervention in the form of sedation or general anesthesia (GA). The choice of anesthetic technique is often guided by individual patient factors and personal clinician practice (Dhakal, Diaz-Gomez, & Freeman, 2015). Two recent meta-analyses (Brinjikji et al., 2015) have found an association of better functional outcome related to endovascular procedures performed under sedation compared to general anesthesia. The interpretation of current data is challenging as most studies are retrospective and performed under direction of non-anesthetists with poor definition of anesthetic techniques. A prospective controlled randomized trial is required to demonstrate the influence of anesthesia techniques on functional outcome. Prior to commencing this large trial, the investigators will execute a feasibility study (GASTROKE-pilot), which is outlined here. Following confirmation of feasibility, the full prospective randomized controlled trial will take place using the same study methodology.

The objectives of the pilot study are: 1) To determine feasibility of the methods and procedures for a proposed prospective randomized controlled trial. Specifically, to determine if randomization can be reliably performed in a timely fashion to facilitate inclusion in the study. Note: EVT will not be delayed beyond institutional temporal limits to allow recruitment or randomization of potential participants. 2) To determine if anesthesia for EVT can be reliably delivered according to the standardized protocol. 3) To determine if post-treatment follow-up of functional outcome can be reliably performed according to a standardized methodology. If the pilot study demonstrates feasibility, the investigators will proceed with a much larger RCT.

Methodology: Randomization: Patients identified by the Acute Stroke team as candidates for EVT will be referred to the study anesthesia team for consideration as study participants. Only after anesthetic pre-procedural assessment is complete, as per usual standard of care, and clinical uncertainty exists as to the best anesthetic management will the patient be randomized. Sequence generation: Randomization will be performed using REDCap to allow central randomization from any hospital computer with internet access. The blocked randomization sequence list will be created in STATA. The randomization instrument will be created in REDCap separate to the data collection tool to ensure blinding allocation is maintained. All treating consultant anesthetists will have access to the REDCap randomization instrument. User rights will be set so that these clinicians do not have access to participant follow-up data. Details of each procedure (GA or sedation) are outlined below. The attending anesthetist will log-on to REDCap and access the Randomization tool. This process will take 2-3 minutes once trained in the randomization process.

Blinding: Both patient and treating physician will be aware of the treatment assignment. Post-procedural functional outcomes will be performed by a dedicated clinician blinded to the treatment assignment. Interventions: Physiological Parameters: Target Values (Talke et al., 2014) • Oxygenation: Maintain SpO2 > 92% and PaO2 > 60 mmHg. • Ventilation: Maintain normocapnia, PaCO2 35-45 mmHg under GA. Avoid respiratory-induced hypercarbia during sedation • Hemodynamics: Systolic blood pressure > 140 mmHg and < 180 mmHg. Diastolic blood pressure < 105 mmHg. • Temperature: Maintain normothermia, T 35°C - 37°C. • Glucose control: Maintain blood glucose concentration 4.0 - 8.0 mmol/L. If blood glucose levels greater than 8 mmol/L (140 mg/dL) IV insulin infusion to be commenced. Blood glucose concentration to be repeated after 30 minutes. Hypoglycemia as defined by blood glucose < 3 mmol/L (50 mg/dL) should be treated with IV 10-20% glucose. General Anesthesia Protocol: (Melinda J. Davis, Cynthia R. Campos-Herrera, & David P. Archer, 2012; Powers et al., 2015; Talke et al., 2014) 1. Monitoring • American Society of Anesthesiologists (ASA) standard (non-invasive blood pressure (BP), electrocardiogram (ECG), oxygen saturation (SpO2), end-tidal carbon dioxide (ETCO2), temperature and neuromuscular monitoring (NMM)) • Invasive BP: direct measure of the arterial BP, with continuous pressure transduction and waveform display is the standard for blood pressure monitoring in AIS. It allows continuous BP assessment and provides reliable vascular access for frequent sampling. However, benefits of invasive arterial monitoring are null if the procedure itself delays reperfusion therapy (Saver, 2006). There is no consensus regarding timing of arterial access in EVT for AIS. This is our protocol: • 1 attempt with the patient awake • Maximum of 2 more attempts with the patient under anesthesia • Stop after a total of 3 attempts, or when the radiologist has access to the femoral artery. 2. Induction of anesthesia. 3. Neuromuscular paralysis. 4. Endotracheal intubation. 5. Positive pressure ventilation: ETCO2 range: 35-40 mmHg until arterial partial pressure of carbon dioxide (PaCO2) is obtained and the gap is measured. 6. Volatile anesthesia with sevoflurane or desflurane to a target age-compensated minimum alveolar concentration (MAC) > 0.5 but = 1(Sivasankar et al., 2016) 7. Vasopressor support: If the systolic BP decreases more than 20% from pre-anesthetic value or is lower than 140 mmHg, the patient will receive vasopressor support as IV phenylephrine and/or ephedrine, titrated to effect. 8. Hypertension management: For systolic BP > 180 mmHg, IV labetalol will be administered, titrated to effect. 9. Arterial blood gas sampling to be performed at the earliest convenience after induction of anesthesia. Clinical goals are outlined above. 10. Temperature monitoring wit esophageal temperature probe. 11. Antagonism of neuromuscular blockade at the end of the procedure. The train of four should be = 0.9 prior to extubation (Hassan et al., 2012; Murphy GS, 2015). 12. Transfer the patient to the post-anesthesia care unit (PACU). Sedation Protocol: 1. Monitoring • ASA standard (non-invasive BP, ECG, SpO2, T, respiratory rate (RR), and ETCO2) • Invasive BP: a direct measure of the arterial blood pressure, • Maximum 3 attempts. Stop after a total of 3 attempts, or when the radiologist has access to the femoral artery. 2. Administer oxygen by nasal prongs or facial mask to achieve a target Sp02 = 92%. 3. Commence sedation: Remifentanil: 0.01-0.06 micrograms/kilogram/minute, titrated to effect. (Janssen et al., 2016) 4. Monitor RR. Decrease sedative infusion rate if RR < 6. 5. Vasopressor support: If the systolic BP decreases more than 20% from pre-anesthetic value or if is lower than 140 mmHg, the patient will receive vasopressor support as IV phenylephrine and/or ephedrine, titrated to effect. 6. Hypertension management: For systolic BP > 180 mmHg, IV labetalol will be administered, titrated to effect. 7. Arterial blood gas sampling to be performed at the earliest convenience after induction of anesthesia. Clinical goals are outlined above. 8. Temperature monitoring with axillary temperature probe. 9. Transfer the patient to the PACU.

Conversion of sedation to GA: Patients randomized to receive EVT under sedation will be converted to GA in cases of emergency (vascular injury), reduced level of consciousness (GCS<8), loss of airway reflexed, respiratory failure with rise in EtCO2 and agitation precluding safe conduct of EVT.

Post-Procedural Follow-up:This will be conducted by a clinical research assistant who is blinded to the study intervention. The specifics of the follow-up procedure are detailed below: Day1: The NIHSS clinical scoring tool will be performed on the stoke inpatient unit. This scale is a validated tool to objectively quantify disability following a stroke. The tool entails assessment of level of consciousness, motor function, sensation, coordination, speech and concentration. Currently, this tool is utilised at LHSC as part of the follow-up for AIS post-procedural days 1. Day 1-2: All patients will have a CT angiogram and MRI within 24-48 hours post-procedure as per usual standard of care. From these scans, the Thrombolysis in Cerebral Infarction (TICI) scale and final infarct volume will be calculated. Day 7: The NIHSS will be repeated to quantify ongoing disability. Day 90: As per the usual standard of care, all patient discharged from hospital will have a 3 month post-stroke outpatient follow-up appointment. The mRS and NIHSS will be repeated by the clinical research assistant at the neurological outpatient appointment. Should the appointment be delayed longer than 3 months post-stroke, a telephone call will be made by the clinical research assistant to determine the mRS. If the patient remains an inpatient at 90 days post-stroke, the electronic record will be accessed to gain the required information to calculate the mRS

ELIGIBILITY:
Inclusion Criteria: All patients with ischemic stroke who:

* are greater than 18 years of age
* considered to be a candidate for endovascular therapy by the London Health Sciences Stroke team
* presenting within the first 8 hours after symptom onset EXCEPT THOSE for whom general anesthesia is thought to be clearly indicated or contraindicated, by the attending anesthesiologist.

Exclusion Criteria:

* Patients in whom the attending anesthesiologist considered that there was a clear indication for either GA or sedation

Ages: 19 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-31 (Estimated); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-08-01 (Estimated)

PRIMARY OUTCOMES:
Randomization potential | 20 weeks
  Total number of participants that have been recruited and the drop out rates. Recruitment goal is 20 patients within 20 weeks.

SECONDARY OUTCOMES:
Number of participants that complete the recruitment procedure prior to start of endovascular treatment. | 20 weeks
  These procedures include patient identification and baseline assessments such as patient co-morbidities, demographics, and pre-procedural anesthetic assessment.
Length of time to complete/completeness of study-related assessments | 1 year
  To assess the feasibility of obtaining completed follow up assessments with this patient population and the time it takes to accomplish this.

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Arango, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Avitsian R, Machado SB. Anesthesia for Endovascular Approaches to Acute Ischemic Stroke. Anesthesiol Clin. 2016 Sep;34(3):497-509. doi: 10.1016/j.anclin.2016.04.004. PMID 27521194
- [Background] Brinjikji W, Murad MH, Rabinstein AA, Cloft HJ, Lanzino G, Kallmes DF. Conscious sedation versus general anesthesia during endovascular acute ischemic stroke treatment: a systematic review and meta-analysis. AJNR Am J Neuroradiol. 2015 Mar;36(3):525-9. doi: 10.3174/ajnr.A4159. Epub 2014 Nov 13. PMID 25395655
- [Background] Dhakal LP, Diaz-Gomez JL, Freeman WD. Role of anesthesia for endovascular treatment of ischemic stroke: do we need neurophysiological monitoring? Stroke. 2015 Jun;46(6):1748-54. doi: 10.1161/STROKEAHA.115.008223. Epub 2015 May 7. No abstract available. PMID 25953376
- [Background] Davis MJ, Menon BK, Baghirzada LB, Campos-Herrera CR, Goyal M, Hill MD, Archer DP; Calgary Stroke Program. Anesthetic management and outcome in patients during endovascular therapy for acute stroke. Anesthesiology. 2012 Feb;116(2):396-405. doi: 10.1097/ALN.0b013e318242a5d2. PMID 22222475
- [Background] Talke PO, Sharma D, Heyer EJ, Bergese SD, Blackham KA, Stevens RD. Republished: Society for Neuroscience in Anesthesiology and Critical Care expert consensus statement: Anesthetic management of endovascular treatment for acute ischemic stroke. Stroke. 2014 Aug;45(8):e138-50. doi: 10.1161/STROKEAHA.113.003412. PMID 25070964
- [Background] Janssen H, Buchholz G, Killer M, Ertl L, Bruckmann H, Lutz J. General Anesthesia Versus Conscious Sedation in Acute Stroke Treatment: The Importance of Head Immobilization. Cardiovasc Intervent Radiol. 2016 Sep;39(9):1239-44. doi: 10.1007/s00270-016-1411-5. Epub 2016 Jul 7. PMID 27387186
- [Background] Sivasankar C, Stiefel M, Miano TA, Kositratna G, Yandrawatthana S, Hurst R, Kofke WA. Anesthetic variation and potential impact of anesthetics used during endovascular management of acute ischemic stroke. J Neurointerv Surg. 2016 Nov;8(11):1101-1106. doi: 10.1136/neurintsurg-2015-011998. Epub 2015 Nov 27. PMID 26614493
- [Derived] Tosello R, Riera R, Tosello G, Clezar CN, Amorim JE, Vasconcelos V, Joao BB, Flumignan RL. Type of anaesthesia for acute ischaemic stroke endovascular treatment. Cochrane Database Syst Rev. 2022 Jul 20;7(7):CD013690. doi: 10.1002/14651858.CD013690.pub2. PMID 35857365